CLINICAL TRIAL: NCT00802880
Title: Determination of Tumor Response Rate by RECIST and FDG-PET Criteria to Dacarbazine in Metastatic Soft Tissue and Bone Sarcoma
Brief Title: Dacarbazine for Metastatic Soft Tissue and Bone Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-1299 / 201109179
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dacarbazine (Experimental): Dacarbazine 850 mg/m^2 IV Day 1 of each 21 day cycle.
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Dacarbazine
  Other Names: DTIC; DTIC-Dome; DIC

SUMMARY:
The purpose of this study is to determine the overall best tumor response rate to dacarbazine given until disease progression as assessed by RECIST criteria, CT and clinical exams in patients with metastatic sarcomas.

DETAILED DESCRIPTION:
The two reasons why dacarbazine was eliminated from treatment options for patients with metastatic sarcoma included inability to effectively address the drug's major toxicities (emesis and neutropenia) and the prevailing opinion that the drug was less effective than other chemotherapeutic agents.

Specific Aim #1: The primary endpoint of this study is to determine the overall best tumor anatomic response rate (CR- complete response, PR - partial response, SD - stable disease, or PD - progressive disease) to dacarbazine given until disease progression as assessed by RECIST criteria using CT and clinical examination in patients with metastatic sarcoma.

The prevailing opinion that dacarbazine was less effective than other chemotherapeutic agents in this setting was not based on data from controlled randomized clinical trials. Indeed, we are not aware of a single randomized trial that was conducted and reported which compared the anti-tumor activity of single agent dacarbazine to that of other active single agents in this patient population. However, phase two trials clearly established that dacarbazine had anti-tumor activity in the treatment of metastatic sarcoma, and our personal experience at this institution has confirmed that this is true. In addition, randomized trials demonstrated that the addition of dacarbazine to doxorubicin increased tumor response rates over doxorubicin alone.12 The literature supports the conclusion that dacarbazine has anti-tumor activity in the treatment of metastatic sarcoma.

Historically, in most studies, tumor response to dacarbazine was assessed by WHO criteria. However, current assessment of tumor response usually is based on RECIST criteria, which differ from the WHO criteria, as shown:

Studies have not been performed to determine the tumor anatomic response rate of single agent dacarbazine using RECIST criteria. This study will determine the tumor anatomic response rate as assessed by RECIST criteria to dacarbazine in patients with metastatic sarcoma. Modern methods of CT scans will be used to assess tumor response which contrasts with the earlier methods to assess tumor response to dacarbazine used in most of the published reports. These methods included physical examination and conventional X-ray or first generation, lower resolution CT scans. The current methods of radiologic assessment of tumor response are superior to those used over 15 years ago. The latest generation of CT scans more accurately measure and image a tumor mass, which may better assess tumor response to therapy.

Specific Aim #2: To determine the overall risk of nausea/emesis (any grade) and neutropenia (grade 3 or 4) with dacarbazine when given with current antiemetic agents (5-hydroxytryptamine-3 serotonin antagonist, dexamethasone, and aprepitant) and with pegfilgrastim.

Historically, dacarbazine-induced toxicities such as emesis and myelosuppression were common and led to significant dose reductions and delays which could have negatively impacted the drug's anti-tumor activity. When dacarbazine was initially identified as a potentially effective agent for the treatment of sarcoma, the anti-emetic drugs available had limited efficacy. Also, there were no measures available to prevent chemotherapy-induced neutropenia. Today, there are very effective drugs that can prevent and reduce the frequency of both chemotherapy-induced emesis and neutropenia.

Dacarbazine carries the risk of emesis (all grades) of >90% of cases when administered without antiemetics13. A three-drug anti-emetic combination of a 5-hydroxytryptamine-3 serotonin antagonist, dexamethasone, and aprepitant is the current recommendation from ASCO when administering highly emetogenic chemotherapy drugs13. Hesketh, et al reported that the risk of emesis (all grades) following highly emetogenic chemotherapy (cisplatin) and pre-medication with this three drug anti-emetic regimen was 27% compared to a two drug regimen of ondansetron and dexamethasone in which the risk was 48% (p< 0.001)14.

Prior studies showed that the risk of grade 3 or 4 neutropenia following dacarbazine given without granulocyte- colony stimulating factors was 36%15. Granulocyte- colony stimulating factors (pegfilgrastim or neupogen) are effective agents in preventing chemotherapy-induced neutropenia. Crawford, et al showed in a randomized trial that risk of chemotherapy- induced grade four neutropenia was one day with G-CSF compared to six days with placebo15. Subsequent randomized trials showed equivalent efficacy of pegfilgrastim compared with neupogen16. Vogel, et al reported in a phase three double blinded randomized trial of patients with breast cancer receiving docetaxel 100 mg/m2 that pegfilgrastim compared to placebo reduced the incidence of febrile neutropenia ( 1% vs 17%, p< 0.001) and febrile neutropenia-related hospitalization (1% vs 14%, p< 0.001)17.

In this trial, we hypothesize that the implementation of these newer anti-nausea agents (5-hydroxytryptamine-3 serotonin antagonist, dexamethasone, and aprepitant) and granulocyte-colony stimulating factor (pegfilgrastim) as a primary prophylactic strategy will reduce the frequency of dacarbazine-induced nausea/emesis (any grade) and neutropenia (grade 3 or 4).

Specific Aim #3: To compare the SUV at up to three target tumor sites and to determine the overall tumor metabolic response (complete metabolic response, partial metabolic response, stable metabolic disease or progressive metabolic disease (CMR, PMR, SMD, or PMD) as assessed by FDG-PET/CT performed at baseline and then after every three cycles of treatment with dacarbazine.

Studies have not been performed to determine the changes in FDG uptake by PET imaging following dacarbazine in patients with metastatic sarcoma. There is limited published data about changes in FDG uptake by PET imaging following other chemotherapy agents in patients with metastatic sarcoma. However, there is an emerging body of data showing the prognostic impact of early tumor response to targeted agents (imatinib or sunitinib) as assessed by FDG-PET in patients with metastatic GIST18. In this trial, we will determine the tumor metabolic response to dacarbazine as assessed by FDG-PET/CT and correlate this to the tumor anatomic response as assessed by CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of soft tissue or bone sarcoma
* Metastatic or locally recurrent and unresectable sarcoma which progressed after one or more prior chemotherapy regimens (excluding adjuvant chemotherapy).
* At least one measurable tumor lesion (by CT scan) At least one FDG avid (SUV ≥ 3) tumor lesion (by PET/CT) which must have been performed at this institution. At least one of these target lesions must be ≥ 1.5 cm in smallest dimension as measured on the baseline CT
* Age greater than 18 yrs old
* ECOG Performance Status of 0-2
* Baseline ANC ≥ 1000/uL, Hgb ≥ 8 Gr/dL, platelets ≥ 100,000/ dL.
* Baseline serum creatinine </= 2.0 mg/dL
* Baseline serum total bilirubin </= 2.0, AST or ALT < 3x ULN
* No active infection
* Signed Informed Consent by patient or legally authorized representative

Exclusion Criteria:

* Current pregnancy or breast feeding.
* A serious uncontrolled medical disorder that in the opinion of the Investigator would impair the ability of the subject to receive protocol therapy.
* Chemotherapy, radiation therapy, or investigational agents given with the last 21 days.
* Investigational agents given with the last 30 days
* Uncontrolled diabetes mellitus. (Subjects with a fasting blood glucose > 200 at time of PET scanning may need to reschedule to another day after consulting with appropriate physicians.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Van Tine, M.D., Ph.D., Principal Investigator — Washington Univerisity School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Antman K, Crowley J, Balcerzak SP, Rivkin SE, Weiss GR, Elias A, Natale RB, Cooper RM, Barlogie B, Trump DL, et al. An intergroup phase III randomized study of doxorubicin and dacarbazine with or without ifosfamide and mesna in advanced soft tissue and bone sarcomas. J Clin Oncol. 1993 Jul;11(7):1276-85. doi: 10.1200/JCO.1993.11.7.1276. PMID 8315425
- [Background] Gottlieb JA, Benjamin RS, Baker LH, O'Bryan RM, Sinkovics JG, Hoogstraten B, Quagliana JM, Rivkin SE, Bodey GP Sr, Rodriguez V, Blumenschein GR, Saiki JH, Coltman C Jr, Burgess MA, Sullivan P, Thigpen T, Bottomley R, Balcerzak S, Moon TE. Role of DTIC (NSC-45388) in the chemotherapy of sarcomas. Cancer Treat Rep. 1976 Feb;60(2):199-203. PMID 769974
- [Background] Buesa JM, Mouridsen HT, van Oosterom AT, Verweij J, Wagener T, Steward W, Poveda A, Vestlev PM, Thomas D, Sylvester R. High-dose DTIC in advanced soft-tissue sarcomas in the adult. A phase II study of the E.O.R.T.C. Soft Tissue and Bone Sarcoma Group. Ann Oncol. 1991 Apr;2(4):307-9. doi: 10.1093/oxfordjournals.annonc.a057942. PMID 1868027
- [Background] Borden EC, Amato DA, Rosenbaum C, Enterline HT, Shiraki MJ, Creech RH, Lerner HJ, Carbone PP. Randomized comparison of three adriamycin regimens for metastatic soft tissue sarcomas. J Clin Oncol. 1987 Jun;5(6):840-50. doi: 10.1200/JCO.1987.5.6.840. PMID 3585441
- [Background] Choi H, Charnsangavej C, Faria SC, Macapinlac HA, Burgess MA, Patel SR, Chen LL, Podoloff DA, Benjamin RS. Correlation of computed tomography and positron emission tomography in patients with metastatic gastrointestinal stromal tumor treated at a single institution with imatinib mesylate: proposal of new computed tomography response criteria. J Clin Oncol. 2007 May 1;25(13):1753-9. doi: 10.1200/JCO.2006.07.3049. PMID 17470865
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on 03/16/2009 and closed to accrual on 12/15/2014.
Period: Overall Study
Arm/Group | Dacarbazine
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dacarbazine
Number analyzed (Participants) | 80
Age, Continuous [Median (Full Range); unit: years] | 53 [20 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 40
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Best Anatomical Tumor Response
Description: * Complete response (CR): disappearance of all target lesions, disappearance of all non-target lesions, normalization of tumor level marker
  * Partial response (PR): at least 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD, persistence of one or more non-target lesion and/or maintenance of tumor marker level above the upper limits of normal
  * Stable disease (SD): neither sufficient shrinkage in target lesions to qualify for PR nor sufficient increase to qualify for progressive disease taking as references the smallest sum LD since the treatment started, persistence of one or more non-target lesion and/or maintenance of tumor marker level above the normal limits of normal
  * Progressive disease (PD): at least 20% increase in the sum of the LD of target lesions and/or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: After completion of 3 cycles
Population: 3 patients failed to complete 3 cycles of treatment due to toxicity. 22 patients failed to complete 3 cycles of treatment due to progressive disease. 1 patient only had PET scan.
Measure: Number; unit: participants
Arm/Group | Dacarbazine
Number analyzed (Participants) | 54
participants
  Complete response | 0
  Partial response | 2
  Stable disease | 22
  Progressive disease | 30

2. Secondary Outcome: Rate of Neutropenia (Grade 3/4)
Description: * Grade 3 neutropenia = absolute neutrophil count of <1000 - 500/mm^3
  * Grade 4 neutropenia = absolute neutrophil count of <500/mm^3
Time Frame: Completion of 6 cycles of treatment (18 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Dacarbazine
Number analyzed (Participants) | 80
percentage of participants | 7.5

3. Secondary Outcome: Rate of Nausea/Emesis (Any Grade)
Description: Approximately 18 weeks
Time Frame: Completion of 6 cycles of treatment (18 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Dacarbazine
Number analyzed (Participants) | 80
percentage of participants | 22.5

4. Secondary Outcome: Comparison of the SUV at up to 3 Tumor Sites
Time Frame: Baseline and after every three cycles of treatment (up to 1 year)
Population: The lower confidence limit is 85% and the upper confidence limit is 95%. 51 patients evaluable at baseline, 50 patients evaluable at end of cycle 3, 20 patients evaluable at end of cycle 6, 7 patients evaluable at end of cycle 9, and 5 patients evaluable at end of cycle 12.
Measure: Mean (95% Confidence Interval); unit: standard uptake value
Arm/Group | Dacarbazine
Number analyzed (Participants) | 51
standard uptake value
  Baseline | 7.42 [6.2 to 8.83]
  End of cycle 3 | 7.57 [6.34 to 9.01]
  End of cycle 6 | 7.7 [6.33 to 9.34]
  End of cycle 9 | 6.89 [5.39 to 8.74]
  End of cycle 12 | 7.48 [5.68 to 9.76]

5. Secondary Outcome: Overall Tumor Metabolic Response
Description: * Complete metabolic response (CMR)-complete resolution of all metabolically active target and non-target lesions, and no interval development of new lesions.
  * Partial metabolic response (PMR)
    * Target lesions: 20% or greater decrease in maximum SUV from baseline. No unequivocal metabolic progression of non-target disease, and no unequivocal new lesions.
    * Non-target lesions: decrease in total number of non-target lesions, without complete resolution of metabolically active disease, or unequivocal decrease in degree of FDG activity within >50% of the lesions. No unequivocal new lesions.
  * Stable metabolic disease (SMD): does not qualify for CMR, PMR, or PMD.
  * Progressive metabolic disease (PMD):
    * Unequivocal development of one more new metabolically active lesions
    * Target lesion: 20% or greater increase in maximum SUV from baseline.
    * Non-target lesions: unequivocal increase in FDG activity
Time Frame: After completion of 3 cycles
Population: 29 patients were not evaluable due to various reasons such as toxicity, progressive disease prior to completion of cycle 3, patient refusal, and no target lesions on PET scan.
Measure: Number; unit: participants
Arm/Group | Dacarbazine
Number analyzed (Participants) | 51
participants
  CMR | 0
  PMR | 4
  SMD | 13
  PMD | 34

6. Secondary Outcome: Correlate the Tumor Metabolic Response Rate With the Tumor Anatomic Response Rate
Time Frame: After completion of 3 cycles
Population: 31 patients were not evaluable due to various reasons such as toxicity, progressive disease prior to completion of cycle 3, patient refusal, and no target lesions on PET scan.
Measure: Number; unit: participants
Arm/Group | Partial Metabolic Response | Stable Metabolic Disease | Progressive Metabolic Disease | Total
Number analyzed (Participants) | 4 | 12 | 33 | 49
participants
  PR | 1 | 0 | 1 | 2
  SD | 2 | 10 | 8 | 20
  PD | 1 | 2 | 24 | 27
  Total | 4 | 12 | 33 | 49

7. Secondary Outcome: Overall Disease Control Rate
Time Frame: 12 months
Population: Only 6 patients were evaluable for response at the end of 12 cycles.
Measure: Number; unit: participants
Arm/Group | Dacarbazine
Number analyzed (Participants) | 6
participants
  Complete response | 0
  Partial response | 0
  Stable disease | 5
  Progressive disease | 1

8. Secondary Outcome: Time to Progression (TTP)
Description: -Progression - At least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Until completion of follow-up (estimated to be 1 year)
Population: 10 patient observations with invalid time or censoring values were not included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine
Number analyzed (Participants) | 70
months | 2.07 [1.84 to 2.30]

9. Secondary Outcome: Overall Survival
Time Frame: Until completion of follow-up or patient death (estimated to be 1 year)
Population: One patient with invalid time or censoring value was not included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine
Number analyzed (Participants) | 79
months | 8.09 [5.56 to 9.74]

10. Secondary Outcome: Correlate the Time to Progression With Best Anatomic Response
Description: as for outcome 8
Time Frame: Completion of follow-up (estimated to be 1 year)
Population: 29 patients were not evaluable due to various reasons such as toxicity, progressive disease prior to completion of cycle 3, patient refusal, and no anatomic response recorded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine
Number analyzed (Participants) | 51
months
  Partial response | NA [9.41 to NA] — The median and upper confidence level were not estimable due to the limited number of events.
  Stable disease | 4.14 [3.91 to 6.94]
  Progressive disease | 1.97 [1.84 to 2.07]

11. Secondary Outcome: Correlate Time to Progression With Best Metabolic Response
Description: as for outcome 8
Time Frame: Completion of follow-up (estimated to be 1 year)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine
Number analyzed (Participants) | 49
months
  Partial metabolic response | 3.95 [1.61 to NA] — The upper confidence level was not estimable due to the limited number of events.
  Stable metabolic disease | 5.30 [2.53 to 9.41]
  Progressive metabolic disease | 2.07 [1.84 to 2.30]

12. Secondary Outcome: Correlate Overall Survival With Best Anatomic Response
Time Frame: Completion of follow-up (estimated to be 1 year)
Population: 26 patients were not evaluable for this outcome measure for various reasons including unknown survival status, progressive disease prior to cycle 3, no anatomic response noted, and toxicity.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine
Number analyzed (Participants) | 54
months
  Partial response | 18.16 [NA to NA] — The lower and upper confidence levels were not estimable due to the limited number of events. Only two patients had partial response and only one of them died within the time frame of the study.
  Stable disease | 14.77 [8.75 to 23.85]
  Progressive disease | 7.96 [5.72 to 10.46]

13. Secondary Outcome: Correlate Overall Survival With Best Metabolic Response
Time Frame: Completion of follow-up (estimated to be 1 year)
Population: 28 patients were not evaluable for this outcome measure due to various reason such as progressive disease prior to cycle 3, unknown survival status, no target lesion on PET scan, and toxicity.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine
Number analyzed (Participants) | 52
months
  Partial metabolic response | 18.16 [7.3 to 25.79]
  Stable metabolic disease | 18.59 [6.91 to 44.01]
  Progressive metabolic disease | 8.75 [6.05 to 12.80]

ADVERSE EVENTS:
Arm/Group | Dacarbazine
Serious Adverse Events (participants affected / at risk) | 16/80
Other Adverse Events (participants affected / at risk) | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacarbazine (N=80)
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Disease progression (General disorders) | 1
Death (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Lung hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Neuropathy - motor (Nervous system disorders) | 1
Abdominal hemorrhage (Gastrointestinal disorders) | 1
Thrombocytopenia (Investigations) | 1
Hypotension (Vascular disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Allergic reaction (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacarbazine (N=80)
Abodominal pain (Gastrointestinal disorders) | 9
Acidosis (Metabolism and nutrition disorders) | 1
Acneiform rash (Skin and subcutaneous tissue disorders) | 1
Albumin - low (Metabolism and nutrition disorders) | 27
Alkaline phosphatase (Investigations) | 19
Allergic reaction/hypersensitivity (Immune system disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anisocoria (Eye disorders) | 1
Anorexia (Gastrointestinal disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bilirubin (Investigations) | 4
Bloating (Gastrointestinal disorders) | 1
Boil (Infections and infestations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 23
Brachycardia (Cardiac disorders) | 1
Bronchospasm: wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Calcium - high (Metabolism and nutrition disorders) | 2
Calcium - low (Metabolism and nutrition disorders) | 29
Chest pain (Cardiac disorders) | 5
Chills (General disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Cold sore (General disorders) | 1
Confusion (Psychiatric disorders) | 2
Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Constipation (Gastrointestinal disorders) | 19
Contracture (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Creatinine (Investigations) | 11
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Diaphoresis (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 13
Disease pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17
Dizziness (Nervous system disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Edema (General disorders) | 22
Elevated PTT (Investigations) | 6
Elevated troponin I (Investigations) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Esophageal obstruction (Gastrointestinal disorders) | 1
Extremity pain (Musculoskeletal and connective tissue disorders) | 3
Face pain (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 43
Fever (General disorders) | 5
Flatulence (Gastrointestinal disorders) | 2
Floaters (Eye disorders) | 1
Flu like syndrome (General disorders) | 2
Frothy urine (Renal and urinary disorders) | 1
GI abdominal hemorrhage (Gastrointestinal disorders) | 3
Glucose - high (Metabolism and nutrition disorders) | 22
Glucose - low (Metabolism and nutrition disorders) | 5
Gout (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 4
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 57
Hot flashes (Vascular disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 5
Hypertriglyceridemia (Investigations) | 1
INR (Investigations) | 9
Inferior vena cava thrombus (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 6
Intraspinal hematoma (Musculoskeletal and connective tissue disorders) | 1
Keratitis (Eye disorders) | 1
Leukocytes (WBC) (Investigations) | 24
Lymphopenia (Investigations) | 54
Memory impairment (Nervous system disorders) | 1
Mood alteration - agitation (Psychiatric disorders) | 1
Mood alteration - anxiety (Psychiatric disorders) | 3
Mucositis (Gastrointestinal disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 18
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathy (sensory) (Nervous system disorders) | 7
Neutropenic fever (Infections and infestations) | 1
Neutrophils (ANC) (Investigations) | 15
Nose hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 1
Phosphorus - low (Metabolism and nutrition disorders) | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 2
Platelets (Investigations) | 33
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pnemonia (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Portal vein thrombosis (Vascular disorders) | 1
Potassium - high (Metabolism and nutrition disorders) | 4
Potassium - low (Metabolism and nutrition disorders) | 12
Proteinuria (Renal and urinary disorders) | 2
Pulmonary embolism (Vascular disorders) | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 4
Reflux gastritis (Gastrointestinal disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
SGOT (AST) (Investigations) | 16
SGPT (ALT) (Investigations) | 15
Seizure (Nervous system disorders) | 3
Shoulder/back pain (Musculoskeletal and connective tissue disorders) | 4
Sinusitis (Infections and infestations) | 1
Sodium - high (Metabolism and nutrition disorders) | 6
Sodium - low (Metabolism and nutrition disorders) | 21
Speech impairment (Nervous system disorders) | 1
Swelling - face (General disorders) | 1
Tachycardia (Cardiac disorders) | 5
Taste alterations (Gastrointestinal disorders) | 3
Thrush (Infections and infestations) | 1
Ulcer: GI duodenum (Gastrointestinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 5
Urinary frequency/urgency (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 5
Urine color change (Renal and urinary disorders) | 1
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Weight loss (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes